CLINICAL TRIAL: NCT01187628
Title: An Open-label, Long-term Extension Study of Lanthanum Carbonate 750 to 2,250 mg in Hyperphosphatemia in Patients With Chronic Kidney Disease Not on Dialysis (52 Weeks Extension From Study 14817)
Brief Title: Long-term Study in Chronic Kidney Disease (Extension From Study 14817)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15074
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Hyperphosphatemia
Keywords: Long-term study in Chronic Kidney Disease; Lanthanum Carbonate
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Fosrenol (Lanthanum Carbonate, BAY77-1931)

INTERVENTIONS:
Drug: Fosrenol (Lanthanum Carbonate, BAY77-1931) — Daily dose: 750-2250mg/day,(270-750mg each 3 times a day) for 52 weeks.

SUMMARY:
The objective of this study is to investigate the safety and the effect on reduction of serum phosphate of long-term administration of lanthanum carbonate (BAY77-1931) 750 to 2250 mg in patients with hyperphosphatemia who completed the 8 week double-blind treatment period of Study 14817 and are judged to be eligible for the long-term extension study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the 8-week double-blind treatment period of Study 14817 and are judged to be eligible for the long-term extension study by the investigator (including those who plan to be on dialysis during the long-term extension study).

Exclusion Criteria:

* Patients with any other conditions that the investigator defines as not appropriate to be enrolled in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | baseline to Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (31):
- Japan (31):
  - Anjo, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Toyohashi, Aichi-ken
  - Yatomi, Aichi-ken
  - Kamogawa, Chiba
  - Kisarazu, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Kyoto, Kyoto
  - Beppu, Oita Prefecture
  - Ōita, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Sakai, Osaka
  - Saga, Saga-ken
  - Shizuoka, Shizuoka
  - Tokushima, Tokushima
  - Koto, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Shinagawa, Tokyo
  - Wakayama, Wakayama